CLINICAL TRIAL: NCT01981759
Title: D-Cycloserine Augmentation of Cognitive Behavioral Therapy for Delusions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-02991
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Delusional Disorder
Keywords: Schizophrenia; Delusions; D-Cycloserine; CBT
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid; Delusions | interventions — Cycloserine; Sugars; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants receive a weekly dose of placebo by mouth one hour before Cognitive Behavioral Therapy (CBT) sessions from week 1-12 (12 visits).
  Interventions: Other: Placebo; Behavioral: Cognitive Behavioral Therapy
- D-Cycloserine (Experimental): Participants will receive a weekly dose of placebo by mouth one hour before Cognitive Behavioral Therapy (CBT) sessions from weeks 1-2 (2 visits), then a weekly 50 mg dose of D-Cycloserine by mouth one hour before CBT sessions from weeks 3-12 (10 visits).
  Interventions: Drug: D-Cycloserine; Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: D-Cycloserine — Participants will receive 10 administrations of 50 mg of D-Cycloserine by mouth one hour before CBT sessions, weekly, in weeks 3-12.
  Other Names: Seromycin
  Arms: D-Cycloserine
Other: Placebo — Participants will receive 12 weekly administrations of placebo by mouth 1 hour before CBT sessions, from weeks 1-12.
  Other Names: Sugar pill
  Arms: Placebo
Behavioral: Cognitive Behavioral Therapy — Participants will engage in a Cognitive Behavioral Therapy treatment plan designed for psychotic delusions. The program will consist of 12 one hour sessions, once weekly from study week 1-week 12.
  Other Names: CBT

SUMMARY:
This study is a placebo-controlled 12 week trial of DCS augmentation of once-weekly CBT sessions in 60 schizophrenia subjects with antipsychotic-resistant delusions. In addition to testing efficacy, this trial will characterize DCS effects in terms of time course and persistence of response and will examine DCS effects on memory consolidation and cognitive flexibility as possible mediators of DCS enhancement of CBT for delusions.

DETAILED DESCRIPTION:
This study consists of a placebo-controlled 12 week trial of DCS augmentation of once-weekly CBT sessions in 60 schizophrenia subjects with antipsychotic-resistant delusions. In addition to testing efficacy, this trial will characterize DCS effects in terms of time course and persistence of response and will examine DCS effects on memory consolidation and cognitive flexibility as possible mediators of DCS enhancement of CBT for delusions. This study will be conducted by the Schizophrenia Research Group of the NYU Langone Medical Center at One Park Avenue 8th Floor and the Psychiatry Outpatient Clinic of Bellevue Hospital located in New York, NY.

Upon signing consent, patients will undergo screening procedures to assess eligibility. A diagnosis of schizophrenia, schizoaffective disorder, or delusional disorder will be determined by the Structured Clinical Interview for DSM IV (SCID) completed by a research clinician using all available clinical data and will be confirmed by consensus diagnosis. A comprehensive medical history and physical exam, including measurement of vital signs, will be performed. A psychiatric history, including diagnosis, treatment history, current medications, and substance use will also be performed. A research assistant will complete the demographics and administer the Scale for Assessment of Positive Symptoms-Delusions (SAPS-D).

At screening only, a fasting blood sample will be obtained to perform routine laboratory tests including electrolytes, BUN, creatinine, liver function tests, fasting glucose, calcium, phosphate, magnesium, albumin and CBC with differential. Urinalysis will be performed to identify unstable medical illness. A urine toxicology screen will be performed and a urine pregnancy test will be done for women of child bearing potential.

Subjects who meet study eligibility criteria will complete the Logical Memory Test portion of the Weschler Memory Scale-III (WMS-III) one week before the baseline visit.

The baseline visit will include the following assessments: SAPS-D, Psychotic Symptom Rating Scales (PSYRATS), Brief Psychiatric Rating Scale (BPRS), Scale for the Assessment of Negative Symptoms (SANS), Calgary Depression Rating Scale (CDRS), Clinical Global Impression (CGI), Heinrich's Quality of Life Scale (Heinrich's QOL), Peter's Delusion Inventory (PDI), Birchwood Insight Scale (BIS), Drug and Alcohol Questionnaire (DAUQ), and the Pittsburg Sleep Quality Index (PSQI) . At the baseline visit the following cognitive assessments will be administered: the Logical Memory Test of the WMS-III, The Wisconsin Card Sort Test (WCST), Verbal Fluency Test (VFT), and the MATRICS Consensus Cognitive Battery (MCCB).

The clinical battery of assessments including the PSYRATS, BPRS, SANS, CDRS, CGI, and Heinrich's QOL will be performed on weeks 4, 8, 12, 24, and 36. The delusions section only of the PSYRATS will be performed on weeks 2, 3, 6, and 10. The Logical Memory Test will be administered on screening visit 2, baseline, week 3, and week 4. The Alternative Beliefs Exercise will occur on weeks 3, 4, and 12. The WCST and VFT will be given to participants at the baseline visit and week 12. Side effects will be assessed using the Systematic Assessment for Treatment Emergent Events (SAFTEE)on weeks 3, 4, 8, and 12.

Beginning at week 1, participants will engage in hour long sessions of Cognitive Behavioral Therapy for delusions. This treatment course will continue weekly from week 1 until week 12 (12 sessions).

For the first two sessions of CBT during weeks 1 and 2, both the experimental and the placebo group will receive a placebo pill by mouth one hour before CBT sessions. Starting week 2, the placebo and experimental groups will receive their respective drugs one hour before CBT sessions from weeks 3-12 (placebo by mouth to placebo group, 50 mg D-cycloserine by mouth to experimental group).

The primary outcome of interest in the study is the change in PSYRATS Delusions Subscale total score compared to placebo from baseline to week 12. Secondary outcome measures include changes as defined by a 20% reduction in PSYRATS Delusions Subscale total score from baseline after 2 weeks of DCS treatment versus placebo as well changes as defined by maintenance of a 20% or greater reduction in the PSYRATS Delusions Subscale total score from baseline at a 3 and 6 month follow up as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-68
* Diagnosis of schizophrenia, schizoaffective disorder, or delusional disorder
* Treated with any antipsychotic except clozapine for at least 8 weeks or antipsychotic naive for lifetime
* Willing to participate in CBT
* Sufficient proficiency in English to complete assessments
* Score of at least 3 on the SAPS at two assessments, four weeks apart

Exclusion Criteria:

* Current treatment with clozapine
* SSRI treatment
* Active alcohol or other substance abuse within six weeks
* Unstable medical illness
* Pregnant or nursing
* Anemia
* Renal insufficiency

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Goff, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Sheppard Pratt, Baltimore, Maryland
  - New York Langone Medical Center/Bellevue Hospital, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As the screening period lasts up to four weeks before the baseline visit and participants are not randomized until week 3, 59 participants were either screen failures or dropped out before randomization to treatment group.
Period: Overall Study
Arm/Group | Placebo | D-Cycloserine
Started (Screened) | 28 | 30
Baseline (Week 1) | 28 | 30
Randomization (Week 3) | 28 | 30
Completed Week 12 | 22 | 22
Completed (Week 36/All Follow-Up) | 21 | 19
Not Completed | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | D-Cycloserine | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.55 (11.97) | 44.60 (13.26) | 44.82 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 16 | 19 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 25 | 28 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data is reported for all participants who reported "race". Not all participants provided responses for this item.
  Participants
    number analyzed (Participants) | 25 | 25 | 50
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 12 | 9 | 21
    White | 10 | 14 | 24
    More than one race | 3 | 1 | 4
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Psychotic Symptoms Rating Scale-Delusions (PSYRATS-D)
Description: The change in the Delusions subscale total of the Psychotic Symptoms Rating Scale (PSYRATS) from Baseline to Week 12. The Delusions subscale is a composite score of 6 items each rated from 0-4 with 4 indicating more severe symptomology. The Delusions subscale has a possible range of 0-24.
Time Frame: Baseline to Week 12
Population: For week 12 values, only those who completed the week 12 assessments are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | D-Cycloserine
Number analyzed (Participants) | 28 | 30
units on a scale
  Baseline PSYRATS Delusion Subscale Total | 14.26 (5.30) | 11.83 (5.58)
  Week 12 PSYRATS Delusion Subscale Total: number analyzed (Participants) | 22 | 22
  Week 12 PSYRATS Delusion Subscale Total | 12.18 (3.79) | 11.91 (5.26)

2. Secondary Outcome: Change in Logical Memory Test-WMS-III
Description: The Logical Memory Test of the Wechsler Memory Scale is a measure of verbal declarative memory. We are using it to evaluate memory consolidation by analyzing the number of thematic elements recalled after a delay of 7 days. Participants are read two different stories-one at Screening visit #2 and one at Baseline. They are asked to recall specific items and narrative themes after 7 days. Scores range from 0-7, 7 indicating perfect thematic recall, and 0 indicating no thematic elements were remembered and worse thematic recall.
  We hypothesize that improved memory consolidation (assessed with the Logical Memory Test) tested 7 days after the first dose of D-cycloserine will predict improvement of delusional scores measured by the PSYRATS-D.
  The reported outcome (change in Logical Memory Test score) was calculated by subtracting the screening visit 2 score from the baseline score for each participant.
Time Frame: 7 days after Baseline, and 7 days after Screening visit 2
Population: Reported summary statistics are for participants randomized at three weeks. One randomized participant is excluded from these results as they did not complete the Logical Memory Test at the baseline visit.
Measure: Mean (Standard Deviation); unit: Change in a score
Arm/Group | Placebo | D-Cycloserine
Number analyzed (Participants) | 27 | 30
Change in a score | -0.96 (1.32) | -1.03 (1.30)

3. Secondary Outcome: Change in Alternate Beliefs Exercise (ABE)
Description: The Alternate Belief Exercise is a measurement of cognitive flexibility. The scores range from 0-21, and a higher score indicates an increased number of alternative beliefs reported.
  This outcome measurement reports the change in number of alternate beliefs generated from weeks 3 to 4 as a predictor of improvement of the PSYRATS Delusions Subscale total score at 12 weeks. Thus a higher score in this outcome measurement indicates a greater number of alternative beliefs reported at week 4 as compared to week 3. This implies greater cognitive flexibility at week 4 as compared to week 3 directly after drug administration.
Time Frame: Week 3 to Week 4
Population: Two participants were randomized and took medication (placebo or DCS) at week 3, but were lost to follow up between week 3 and week 4. One participant was randomized at week 3 but did not take medication or complete the ABE exercise at week 3. These three participants are not included in the reported data.
Measure: Mean (Standard Deviation); unit: Change in a score
Arm/Group | Placebo | D-Cycloserine
Number analyzed (Participants) | 26 | 29
Change in a score | 1.15 (2.80) | 0.59 (1.84)

ADVERSE EVENTS:
Time Frame: Entire study duration, from Randomization through the final follow-up at Week 36.
Description: Adverse Event reporting is based on self-report on the Systematic Assessment of Treatment Emergent Effects (SAFTEE).
Groups:
- D-Cycloserine: Participants will receive a weekly dose of 50 mg placebo by mouth one hour before Cognitive Behavioral Therapy (CBT) sessions from weeks 1-2 (2 visits), then a weekly 50 mg dose of D-Cycloserine by mouth one hour before CBT sessions from weeks 3-12 (10 visits).
  Cognitive Behavioral Therapy: Participants will engage in a Cognitive Behavioral Therapy treatment plan designed for psychotic delusions. The program will consist of 12 one hour sessions, once weekly from study week 1-week 12.
Arm/Group | Placebo | D-Cycloserine
All-Cause Mortality (participants affected / at risk) | 24/28 | 24/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 3/30
Other Adverse Events (participants affected / at risk) | 24/28 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | D-Cycloserine (N=30)
Psychiatric Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)
Medical Hospitalization (Infections and infestations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | D-Cycloserine (N=30)
Appetite Decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Appetite Increased (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Abdominal Discomfort (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorgasmia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0)
Auditory Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Back Ache (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Blisters (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood Sugar Increased (Endocrine disorders) | 0 (0) | 1 (1)
Blurred Vision (Eye disorders) | 3 (3) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Burning Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chest Pain (Vascular disorders) | 1 (1) | 1 (1)
Common Cold (Infections and infestations) | 4 (5) | 1 (2)
Concentration Impaired (Nervous system disorders) | 0 (0) | 2 (2)
Nasal Congestion (Infections and infestations) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Impaired Coordination (Nervous system disorders) | 1 (1) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Decreased Sleep (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Difficulty Thinking (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness Upon Standing (Nervous system disorders) | 1 (1) | 0 (0)
Drooling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Drowsiness (Nervous system disorders) | 2 (2) | 0 (0)
Drowsy on Awakening (Nervous system disorders) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 2 (2) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ear Feels Clogged (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye Hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Facial Swelling (General disorders) | 1 (1) | 0 (0)
Faintness (Vascular disorders) | 0 (0) | 1 (1)
Falling Down (Nervous system disorders) | 0 (0) | 1 (1)
False Sensation (Nervous system disorders) | 0 (0) | 2 (2)
Fatigue (Nervous system disorders) | 1 (1) | 4 (5)
Feeling Strange (Psychiatric disorders) | 0 (0) | 1 (1)
Flu-like Symptoms (Infections and infestations) | 0 (0) | 1 (1)
Frequency of Urination (Hepatobiliary disorders) | 0 (0) | 2 (2)
Gingival Bleeding (Infections and infestations) | 0 (0) | 1 (1)
Hair Loss (General disorders) | 0 (0) | 1 (1)
Hair Thinning (General disorders) | 1 (2) | 1 (1)
Hallucinations (Psychiatric disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 5 (6)
Hot Flashes (General disorders) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Incarceration (Social circumstances) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 3 (3) | 5 (5)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Libido Decreased (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lung Disease Obstruvtive (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Memory Impaired (Nervous system disorders) | 1 (1) | 2 (2)
Mental Concentration Difficulty (Nervous system disorders) | 0 (0) | 1 (1)
Mental Dullness (Nervous system disorders) | 0 (0) | 1 (1)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscle Spasm/Twitch (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Muscle Weakness/Fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nervousness (Psychiatric disorders) | 0 (0) | 3 (3)
Nightmares (Nervous system disorders) | 2 (3) | 4 (4)
Numbness (Nervous system disorders) | 0 (0) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Pneumonia and Dehydration (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT01981759/Prot_SAP_000.pdf